CLINICAL TRIAL: NCT02205216
Title: Can Transcranial Direct Stimulation Enhance the Efficacy of a Rehabilitative Intervention for the Treatment of Freezing of Gait in Parkinson's Disease? A Double Blind Randomized Controlled Study
Brief Title: Can tDCS Enhance Efficacy of Rehabilitative Intervention for Freezing of Gait in Parkinson's Disease?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, David Benninger, MD, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: VD226/14
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Parkinson Disease
Keywords: tDCS; FOG; Freezing of Gait; Parkinson; Rehabilitation
MeSH Terms: conditions — Parkinson Disease | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (Active Comparator): Active tDCS combined with a rehabilitative intervention consisting of cognitive training and sensory cueing.
  Interventions: Device: Active tDCS; Behavioral: Rehabilitation Therapy
- Sham tDCS (Sham Comparator): Sham tDCS combined with a rehabilitative intervention consisting of cognitive training and sensory cueing.
  Interventions: Device: Sham tDCS; Behavioral: Rehabilitation Therapy

INTERVENTIONS:
Device: Active tDCS — anode over the motor and premotor cortex with cathodes placed over both mastoids. TDCS will be applied for 20 minutes at 2 mA.
  Arms: Active tDCS
Device: Sham tDCS — anode and cathode placed 1 cm apart over the forehead and DC (1mA) applied for 1-2 min, short-circuited through the skin creating the same temporary "tingling" sensation without effects on the brain.
  Arms: Sham tDCS
Behavioral: Rehabilitation Therapy — All patients will undergo a rehabilitation therapy intervention (2x a week for 4 weeks = 8 intervention sessions) with simultaneous sham or active tDCS. The trained physiotherapist will follow a standardized program with checklist. Each of the 8 training session will last approximately 45min. The rehabilitative interventions include:
  1. cognitive training: attentional strategies (mental counting, mental obstacle)
  2. transfer training: everyday activities
  3. motor training (walking) with sensory cueing (visual, acoustic, cane, ball) The rehabilitation therapy is divided into two sessions both including a 5 minutes warm-up and the learning of cueing and movement strategies based on different modalities (cognitive, visual, tactile and auditory).

SUMMARY:
Freezing of gait in Parkinson's disease (PD) is a major cause of disability and falls and responds often incompletely to conventional therapy. The pathogenesis remains largely unknown and therapeutic alternatives are needed. Rehabilitative interventions that consist of learning cognitive strategies with sensory cueing to prevent and to overcome FOG represent the most efficacious intervention, but difficulties in learning and execution of these cognitive strategies are the main cause of failure. Transcranial direct current stimulation (tDCS) enhances motor task learning and execution in patients with PD and might enhance the efficacy of rehabilitative interventions.

This study intends to address the following question whether tDCS can enhance the efficacy of rehabilitative interventions in the treatment of freezing of gait in Parkinson's disease?

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 30 to 80 years with DOPA-responsive PD Hoehn and Yahr (HY) grade of 2 to 4 while "off"
* must be on a regimen including levodopa
* total dose of levodopa and dopamine agonists (using dopamine equivalents) has to be equal to or more than 300 milligrams per day
* Gait difficulties with Freezing of Gait as defined by MDS-UPDRS I score ≥ 2 in FOG
* Optimal conventional PD medication for > 1 month prior to screening
* scheduled for rehabilitative intervention for the treatment of freezing of gait

Exclusion Criteria:

* significant concurrent medical or psychiatric disease
* history of seizures and epilepsy
* Dementia or other neurodegenerative disease (besides PD)
* pallidotomy, implanted electrodes and generator for deep brain stimulation
* pregnancy
* surgically or traumatically implanted foreign bodies such as an implanted medical pump, implanted hearing aids, metal plate in the skull, or metal implant in the skull or eyes (other than dental appliances or fillings) that may pose a physical hazard during tDCS.
* Study would cause undue risk or stress for reasons such as tendency to fall, excessive fatigue, general frailty, or excessive apprehensiveness.
* significant postural instability with daily falls, inability to walk the parcours or inability to walk 10 meters.
* presence of significant cognitive dysfunction as determined by Montreal Cognitive Assessment (MOCA) <20 or mentally impaired patients having no capacity to provide their own consent (the physician establishing the diagnosis and applying UPDRS will evaluate patient's mental capacity using conventional clinical interview).
* presence of other co-morbid conditions that can contribute to gait dysfunction (orthopedic, rheumatologic, cardiac, other)
* presence of clinically significant hallucinations
* participation in any rehabilitation therapy for FOG within the last six months prior to screening

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Walking parcours | from baseline to one month follow-up
  This standardized parcours, performed under guidance of a physiotherapist, includes real-life conditions which are known to precipitate freezing. Time needed to perform the parcours and number of FOG episodes will be assessed.

SECONDARY OUTCOMES:
New Freezing of Gait Questionnaire (N-FOGQ) | from baseline to follow-up periods (immediately, 1 and 3 months after the last intervention)
  NFOG-Q is a widely used and validated questionnaire for quantifying FOG severity and frequency in the daily living
Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | from baseline to follow-up periods (immediately, 1 and 3 months after the last intervention)
39-Item Parkinson's Disease Questionnaire (PDQ-39) | from baseline to follow-up periods (immediately, 1 and 3 months after the last intervention)
Beck Depression Inventory (BDI) | from baseline to follow-up periods (immediately, 1 and 3 months after the last intervention)
10 Meter Walk Test (10MWT) | from baseline to follow-up periods (immediately, 1 and 3 months after the last intervention)
  10MWT measures the time taken and the number of steps needed to walk a 10-meter distance from a standing position. Gait testing includes three averaged trials.
Timed Up & GO (TUG) | from baseline to follow-up periods (immediately, 1 and 3 months after the last intervention)
  TUG requires patients to get up of a standard armed-chair, to walk 3 meters away, to turn around a cone, to walk back and to sit down.

CONTACTS AND LOCATIONS:
Overall Officials: David Benninger, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland